CLINICAL TRIAL: NCT07395180
Title: Differentiation of Human Body Balance Disorders - Analysis of the Potential of Functional Tests in Determining the Cause of Disorders
Brief Title: Differentiation of Human Body Balance Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Anna Olczak, PhD; Senior Specialist of the Rehabilitation Clinic, Military Institute od Medicine National Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 12/KRN/24
Record Dates: First submitted 2026-01-18; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Visual Defects; Labyrinth Diseases; Cervical Spine Degenerative Disease; Healthy; Posterior Columns of the Spinal Cord
Keywords: stroke; posterior columns of the spinal cord; cervical spine degenerative disease; labyrinth diseases; visual defects; healthy; balance
MeSH Terms: conditions — Stroke; Vision Disorders; Labyrinth Diseases

STUDY DESIGN:
Intervention Model Description: . Type of research - study with a control group; Study Group - patients after a stroke/cerebellum, with changes in the posterior cords of the spinal cord, with degenerative changes of the spine, including the cervical section, with labyrinth disorders, with uncorrected vision defects. Control group - healthy volunteers. Age of the respondents - range from 20 to 80 years; women and men, in the acute and subacute period of the disease, as well as healthy volunteers. The group size with a moderate effect (f = 0.25), alpha = 0.05, and test power = 0.95 will be > 324 people (54 people in each group).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Patients after stroke (Experimental)
  Interventions: Diagnostic Test: Patients after stroke; Diagnostic Test: Patients with posterior columns of the spinal cord; Diagnostic Test: Patients with labyrinth diseases; Diagnostic Test: Patients with visual defects; Diagnostic Test: Patients with cervical spine degenerative disease; Diagnostic Test: Healthy participants
- Patients with posterior columns of the spinal cord (Experimental)
  Interventions: Diagnostic Test: Patients after stroke; Diagnostic Test: Patients with posterior columns of the spinal cord; Diagnostic Test: Patients with labyrinth diseases; Diagnostic Test: Patients with visual defects; Diagnostic Test: Patients with cervical spine degenerative disease; Diagnostic Test: Healthy participants
- Patients with labyrinth diseases (Experimental)
  Interventions: Diagnostic Test: Patients after stroke; Diagnostic Test: Patients with posterior columns of the spinal cord; Diagnostic Test: Patients with labyrinth diseases; Diagnostic Test: Patients with visual defects; Diagnostic Test: Patients with cervical spine degenerative disease; Diagnostic Test: Healthy participants
- Patients with visual defects (Experimental)
  Interventions: Diagnostic Test: Patients after stroke; Diagnostic Test: Patients with posterior columns of the spinal cord; Diagnostic Test: Patients with labyrinth diseases; Diagnostic Test: Patients with visual defects; Diagnostic Test: Patients with cervical spine degenerative disease; Diagnostic Test: Healthy participants
- Patients with cervical spine degenerative disease (Experimental)
  Interventions: Diagnostic Test: Patients after stroke; Diagnostic Test: Patients with posterior columns of the spinal cord; Diagnostic Test: Patients with labyrinth diseases; Diagnostic Test: Patients with visual defects; Diagnostic Test: Patients with cervical spine degenerative disease; Diagnostic Test: Healthy participants
- Healthy participants (Other)
  Interventions: Diagnostic Test: Patients after stroke; Diagnostic Test: Patients with posterior columns of the spinal cord; Diagnostic Test: Patients with labyrinth diseases; Diagnostic Test: Patients with visual defects; Diagnostic Test: Patients with cervical spine degenerative disease; Diagnostic Test: Healthy participants

INTERVENTIONS:
Diagnostic Test: Patients after stroke — Body posture assessment (APECS), the Tandem test, the Trunk Stability test, the modified Rankin Scale to assess the general physical impairment of patients, and the National Institute for Health Stroke Scale (NIHSS) to determine the neurological deficit. , and the Modified Ashworth Scale, Romberg test, Fukuda test, differential test for vertigo, Unterberg test, body balance test using Biodex SD balance platform, Cervical spine muscle tone test using Luna EMG.
Diagnostic Test: Patients with posterior columns of the spinal cord — Body posture assessment (APECS), the Tandem test, the Trunk Stability test, the modified Rankin Scale to assess the general physical impairment of patients, and the National Institute for Health Stroke Scale (NIHSS) to determine the neurological deficit. , and the Modified Ashworth Scale, Romberg test, Fukuda test, differential test for vertigo, Unterberg test, body balance test using Biodex SD balance platform, Cervical spine muscle tone test using Luna EMG.
Diagnostic Test: Patients with labyrinth diseases — Body posture assessment (APECS), the Tandem test, the Trunk Stability test, the modified Rankin Scale to assess the general physical impairment of patients, and the National Institute for Health Stroke Scale (NIHSS) to determine the neurological deficit. , and the Modified Ashworth Scale, Romberg test, Fukuda test, differential test for vertigo, Unterberg test, body balance test using Biodex SD balance platform, Cervical spine muscle tone test using Luna EMG.
Diagnostic Test: Patients with visual defects — Body posture assessment (APECS), the Tandem test, the Trunk Stability test, the modified Rankin Scale to assess the general physical impairment of patients, and the National Institute for Health Stroke Scale (NIHSS) to determine the neurological deficit. , and the Modified Ashworth Scale, Romberg test, Fukuda test, differential test for vertigo, Unterberg test, body balance test using Biodex SD balance platform, Cervical spine muscle tone test using Luna EMG.
Diagnostic Test: Patients with cervical spine degenerative disease — Body posture assessment (APECS), the Tandem test, the Trunk Stability test, the modified Rankin Scale to assess the general physical impairment of patients, and the National Institute for Health Stroke Scale (NIHSS) to determine the neurological deficit. , and the Modified Ashworth Scale, Romberg test, Fukuda test, differential test for vertigo, Unterberg test, body balance test using Biodex SD balance platform, Cervical spine muscle tone test using Luna EMG.
Diagnostic Test: Healthy participants — Body posture assessment (APECS), the Tandem test, the Trunk Stability test, the modified Rankin Scale to assess the general physical impairment of patients, and the National Institute for Health Stroke Scale (NIHSS) to determine the neurological deficit. , and the Modified Ashworth Scale, Romberg test, Fukuda test, differential test for vertigo, Unterberg test, body balance test using Biodex SD balance platform, Cervical spine muscle tone test using Luna EMG.

SUMMARY:
Our research aims to analyze the possibilities of functional assessment of imbalances in the human body. Using the available, commonly known and used tests and devices for objective examination of static and dynamic body balance, as well as changes in the tension of selected muscles of the cervical spine in static and dynamic conditions, depending on visual control or its absence, we hope to identify important research tools that help to differentiate the causes of imbalances. Studies conducted on a group of healthy people and groups of patients: after a stroke, with changes in the posterior cords of the spinal cord, with labyrinth disorders, with degenerative changes in the spine, with visual impairments, and in healthy people, seem to be important in the analysis of the discussed topic. The investigators will answer the following detailed research questions: 1. Does the type of disease/disease or its absence affect the human balance in the Romberg test? 2. Do visual defects affect the tension of the muscles of the cervical spine? 3. Do changes in the muscle tension of the cervical spine affect the ability to maintain balance in the Unterberger test? 4. Do the mobility deficits in the cervical spine coincide with cervical or labyrinthine balance disorders in the differential test for vertigo and in the Fukuda test? 5. How does the tension of the muscles of the cervical spine change in the tested groups on the stable and unstable, depending on the vision control? 6. Does the type of disease/illness or its absence affect changes in the tension of the muscles of the cervical spine, and does it correlate with the balance of the body on a stable and unstable surface? The results of the research may facilitate the functional differentiation of imbalances in the human body. The investigators hypothesize that functional tests will help determine the cause of imbalance in the human body. This will allow us to determine with high probability the dominant cause of balance disorders (eye disorders, changes in the cervical spine / musculoskeletal system, labyrinth, proprioceptors, cerebellum, posterior cords of the spinal cord), already at the initial stage of diagnosis. The research will improve the process of implementing effective treatment and therapeutic procedures.

ELIGIBILITY:
Inclusion Criteria:

* 1) stroke patients (7 to 9 weeks after cerebellar stroke), with degenerative changes of the spine, including the cervical section, with labyrinth disorders, with visual defects, with changes in the posterior cords of the spinal cord;
* 2) functional status of patients that allows them to stand and walk in place and over a distance (Rankin ≤ 3);
* 3) Modified Ashworth Muscle Tone Scale (MAS ≤1/1+);
* 4) positive Tandem test;
* 5) no major deficits in communication, memory or comprehension which may impede correct measurement;
* 6) over 20 years of age; maximum 80 years.

The main criteria for inclusion in the control group:

* 1) healthy people with a stable trunk (100 TCT points);
* 2) having normal muscle tone (MAS=0), walking independently;
* 3) at least 20 years old; maximum 80 years.

Exclusion Criteria:

* 1) coexisting diseases considered in the study;
* 2) stroke up to seven weeks after the episode;
* 3) epilepsy;
* 4) lack of trunk stability;
* 5) lack of independent standing and walking;
* 6) high or very low blood pressure, dizziness, malaise.

Criteria for exclusion from the control group:

* 1) history of neurological or musculoskeletal disorders, such as stroke or brain injury, or other neurological conditions that may affect their ability to move the trunk and legs actively;
* 2) degenerative changes, labyrinth disorders, vision defects;
* 3) pain, dizziness;
* 4) constant use of orthopedic supplies;
* 5) severe deficits in communication, memory, or comprehension, which may make it difficult to perform the measurement correctly;
* 6) high or very low blood pressure, feeling unwell.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Advanced Packaging and Heterogeneous Integration for Electronic Components and Systems (APECS) | Day 1
  Evaluation of body posture in the frontal and sagittal planes - Advanced Packaging and Heterogeneous Integration for Electronic Components and Systems (APECS)
The Tandem Test | Day 1
Modified Ashworth Scale (MAS) | Day 1
Trunk Stability Test | Day 1
Rankin Scale | Day 1
NATIONAL INSTITUTES OF HEALTH STROKE SCALE (NIHSS) | Day 1

SECONDARY OUTCOMES:
Romberg test | Day 1
Fukuda test | Day 1
Differential test for vertigo | Day 1
Body balance test on the Biodex SD platform | Day 1
Cervical spine muscle tone test using Luna EMG | Day 1
Unterberger test | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Military Institute od Medicine National Research Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No